CLINICAL TRIAL: NCT02509338
Title: Validation of an Electrode Internal Globus Pallidum Deep Brain Stimulation Lead Implantation for Treatment of Dystonia
Brief Title: Validation of the Implantation of a New Electrode for the Treatment of Dystonia
Acronym: MONOCONTACT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The medical device arrived at expirationand it was not possible to have new one
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9053
Record Dates: First submitted 2015-07-20; First posted 2015-07-28 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Generalized Dystonia; Segmental Dystonia; Tardive Dystonia
MeSH Terms: conditions — Tardive Dyskinesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electrode deep brain stimulation (Experimental): Monocontact electrode deep brain stimulation
  Interventions: Device: Electrode deep brain stimulation (Monopolar DBS Lead Model 09064-40cm)

INTERVENTIONS:
Device: Electrode deep brain stimulation (Monopolar DBS Lead Model 09064-40cm) — Deep brain stimulation surgery with implantation of one contact-electrode deep brain stimulation electrodes bilaterally in the internal globus pallidum for treating dystonia

SUMMARY:
The main objective of the trial is to study the technical feasibility of the implantation of a new electrode Monocontact deep brain stimulation electrode in dystonia.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) is a validated therapy for treating dystonia and other movement disorders. The main therapeutical target used for treating dystonic syndromes is the internal globus pallidum (GPi). Given the morphology and the topography of this nucleus and, based on the experience of an efficient therapy by using only one or two contacts out of the available four contacts of the standard DBS lead, we designed two new electrodes, one one contact-electrode and one two contact-electrodes, with the aim to limit side effects related to internal globus pallidum DBS and to provide a more homogeneous electric field around the electrode within the GPi and maintaining the same therapeutical outcome.

The main objective of the trial is to study the technical feasibility of the implantation of a new one contact-electrode (Monopolar DBS Lead Model 09064-40cm) for treating isolated generalized/segmental dystonia or tardive dystonia.

The second main objective of the study is to assess the safety of the implantation of the new device.

The secondary objective is to explore the therapeutical effect of DBS using the new monocontact electrode and to study the electrical field generated around the monocontact electrode within the GPi.

The study is prospective and patients are recruited from a Tertiary Movement Disorders Clinic. Seven subjects will be recruited for the study.

ELIGIBILITY:
Inclusion Criteria:

* Age superior to 18 years and inferior to 65 years
* Generalized or segmental isolated dystonia or tardive dystonia
* Diagnosis is based on history, clinical examination, check-up without abnormalities and normal brain MRI allowing exclusion of secondary and degenerative dystonias
* Unsufficient response to pharmacological treatment (improvement < 30/% on clinical dystonia scales)
* No comorbidity interfering with general anesthesia, or representing contraindication for neurosurgical procedure or with the follow-up during the trial
* Consent of the patient
* Insurance affiliation
* Follow-up possible for 12 months
* Available insurance for the operated patient

Exclusion Criteria:

* No possibility for clinical follow-up
* Acquired dystonia except for tardive dystonia
* MRI or generalized anesthesia contraindicated
* Anticoagulant treatment or antiaggregant treatment
* Pregnancy
* Ongoing participation to another clinical trial
* Guardianship or Trusteeship
* Person deprived of liberty

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Technical feasibility of new electrode implantation | One year
  The feasibility of the implantation is evaluated by stereotaxic frame placement, site of incision, burr hole size and location, technique for insertion, connection with the extension cables to the neurostimulator, measure of the impedances, duration of the surgery, MRI control for lead position, comparison of the artefacts of the leads with the artefacts of the standard electrodes.
Safety of new electrode implantation (evaluated by the occurence of side effects) | One year
  The safety of the implantation is evaluated by the occurence of side effects after the implatation and along the follow-up.

SECONDARY OUTCOMES:
clinical effect of deep brain stimulation using one contact-electrodes (Burke Fahn Marsden's dystonia rating scale and the Toronto Western Spasmodic Torticollis Rating Scale) | One year
  Clinical change as measured by the decrease of the motor and disability of the patient (Burke Fahn Marsden's dystonia rating scale and the Toronto Western Spasmodic Torticollis Rating Scale).

CONTACTS AND LOCATIONS:
Overall Officials: Laura A CIF, MD, PhD, Principal Investigator — CHRU Montpellier
Locations (1):
- Chru Montpellier, Montpellier, France